CLINICAL TRIAL: NCT05417997
Title: Evaluation of Effects, Safety, Viral Load and Antibody Level of Functional Food Dietary Supplement Containing Grape Products in Controlled, Randomized Study Using SARSCoV-2 RT-PCR Positive Covid-19 Patients.
Brief Title: Effect of Kunamin in SARS-CoV-2 RT-PCR Positive Covid-19 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RAAS Nutritionals, LLC (Industry)
Collaborators: Kayseri City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APRON 2020-OK-01
Record Dates: First submitted 2022-05-18; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Respiratory Infection; FLU; Cold; Influenza; Bacterial Pneumonia; COVID-19 Pneumonia
MeSH Terms: conditions — Common Cold; Influenza, Human; Pneumonia, Bacterial | interventions — favipiravir; Enoxaparin; Lansoprazole; Acetaminophen; Ceftriaxone; Clarithromycin; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: The interventions were assigned to participants based on results of in vitro and in vivo studies on H1N1 virus and efficacy for interventions that were used in the study. Kunamin is a botanical drug containing no toxicity. The intervention contain KH good healthy cells (proteins). The intervention not only treat and cure but also can prevent COVID-19 for those who are infected with COVID-19 only by producing antibodies against COVID-19. Therefore, it can be used as a combined drug and oral vaccine to treat, cure and prevent COVID-19. Just like COVID-19 vaccine, the more interventions patients take, the longer period of protection. The strategy is determined by the principal investigator depending on the severity of the illness. The interventions can help prevent COVID-19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research Arm (Experimental): Kunamin® 20 capsules 500mg daily plus; Standard therapy interventions determined and prescribed by investigators including:
  * Favipiravir: 1,600 mg (8 tablets) by mouth twice daily for 5 days.
  * Enoxaparin: 40 mg SQ daily if D-dimer < 3000 ng/mL *or* plt < 100,000
  * Enoxaparin: 0.5 mg/kg SQ twice daily if D-dimer >3000 ng/mL *and* plt < 100,000
  * Lansoprazole: 30 mg (one tablet) by mouth, once a day for 7 days.
  * Paracetamol: 500 mg (one tablet) by mouth, up to one tablet every 4 to 6 hours in case of fever (100.4°F/38°C or higher).
  * Ceftriaxone: 500 mg IV once a day for 5-7 days.
  * Clarithromycin: 250 mg (one tablet) twice a day for 5-7 days.
  * Methylprednisolone: 80 mg/kg IV bolus, followed by an infusion of 80 mg/day in 240 mL normal saline at 10 mL/h.
  Interventions: Dietary Supplement: Kunamin®; Drug: Favipiravir; Drug: Enoxaparin; Drug: Lansoprazole; Drug: Paracetamol; Drug: Ceftriaxone/ Clarithromycin; Drug: Methylprednisolone
- Control arm (Placebo Comparator): According to MOH of Turkey, which required a standard treatment including the following drugs as placebo:
  * Favipiravir
  * Enoxaparin
  * Enoxaparin
  * Lansoprazole
  * Paracetamol
  * Ceftriaxone/ Clarithromycin
  * Methylprednisolone
  Interventions: Drug: Favipiravir; Drug: Enoxaparin; Drug: Lansoprazole; Drug: Paracetamol; Drug: Ceftriaxone/ Clarithromycin; Drug: Methylprednisolone

INTERVENTIONS:
Dietary Supplement: Kunamin® — Grape juice, seed, stem and rice extracts supplement containing KH good healthy cells (proteins)
  Arms: Research Arm
Drug: Favipiravir — Antiviral medication used to treat influenza
Drug: Enoxaparin — Anticoagulant medication
Drug: Lansoprazole — Treat stomach ulcers, a damaged esophagus, gastroesophageal reflux disease (GERD), and high levels of stomach acid.
Drug: Paracetamol — Analgesic to treat minor aches and pains, and fever reducer.
Drug: Ceftriaxone/ Clarithromycin — Inhibits the production of pneumolysin
Drug: Methylprednisolone — Treat inflammation, severe allergies, flares of chronic illnesses

SUMMARY:
The primary objective of this study is to determine the safety and efficacy profile of the food supplement (KUNAMIN®) containing grape juice, seed, stem, and bark given to patients treated with the established treatment regimen against novel coronavirus infectious disease (COVID-19) via comparing Kunamin® group versus control group in a clinical trial.

In this study, both the therapeutic effect and the safety of the Kunamin® product has been evaluated. The study has been conducted on COVID-19 infected patients. Within the scope of the study, Covid-19 patients consisting of male and female patients are examined to evaluate the therapeutic effect.

COVID-19 infected patients are divided into 2 groups and the treatment group received grape food supplements for 15 days in addition to their standard treatment. The other group received only standard therapy. The effects of supplements containing grape products on the COVID-19 infection process of patients are investigated, as indicated in the primary, secondary, and tertiary endpoints. For this purpose, both the observation of routine examination findings and the effectiveness of food supplements on viral load and antibody levels are investigated. In the follow-up that continues for 30 days, COVID-19 Rapid Antigen test made in USA approved by FDA is used to monitor the efficacy of Kunamin® as patient treated by Kunamin® viral load is diminished either after 5 days, 10 days or 15 days, COVID-19 Rapid Antibody test made in USA approved by FDA has been used to monitor the development of IgM and IgG antibodies on day 0, day 5th, day 10th, day 15th and day 30th in addition to PCR test of Perkinelmer by Kayseri hospital. In conjunction, the sponsor used AIT Laboratories A HealthTrackRx Company PCR test CLIA and FDA approved for not only COVID-19 but also 27 kinds of cold and flu viruses and 90 different kinds of bacteria.

The number of patients planned for randomization was 240, however due to dropouts the hospital was able to screen 132 patients. Out of 132 patients we were able to enroll randomized total of 71 patients, 47 patients in the research arm and 24 in the control arm.

DETAILED DESCRIPTION:
We conducted a medical observation from December 2019 when there were no cases and no deaths in America, and just the revelation of this new disease in China. There is still no cure for COVID-19, a very contagious disease that has a tendency to destroy the immune system and has caused many mysterious complications while vaccination is a long-term strategy.

The complete study involved 100 outpatients from January 2020 to February 2021 who attended our clinic with flu, cold and respiratory symptoms, studied with a panel of 27 viruses and 90 bacteria which has been considered as phase 1 and phase 2 clinical trial for Kunamin® in the United States of America.

The sponsor also contracted with CRO APRON in Turkey to conduct the third phase clinical trial for Kunamin® for COVID-19 inpatients in Kayseri City Hospital. The number of patients planned for randomization was 240, however due to dropouts, we were able to screen 132 patients. Out of these 132 patients, we enrolled a total of 71 patients and randomized 47 patients in the research arm and 24 in the control arm.

The median age for COVID-19 positive patients is 39.6 years old (range of 18-64 years). Forty (56%) are female and 31 (44%) are male. The demographics include all Caucasians.

3 (4%) out of 71 patients after 40 capsules of Kunamin® were admitted into ICU and intubated, 100% survived.

Nineteen (40%) of our patients in the Turkey study had adverse events. Only one patient who completed the 30-day trial experienced an adverse event. 17 volunteers left the trial by their own will because of gastrointestinal tract related adverse events. All the vital signs were in normal ranges in control and treatment group. No serious adverse events or fatality occurred during the trial. We think the problem with the gastrointestinal tract related adverse events is not caused by Kunamin, but by the standard treatment including at least 6 drugs. In USA our medical observation for 100 patients we used only Kunamin and we found only two minor gastrointestinal tract related adverse events (2%), including one overdose of Kunamin in one patient, and the use of antibiotics in another. According to FDA rules and regulations, it is not allowed to mix a botanical drug with a chemical drug, therefore we should never use Kunamin together with standard treatment which consisted of several drugs. The Ministry of Health in Turkey for safety of COVID-19 patients required that Kunamin should be used along with hospital's standard treatment.

Thanks to grape, rice, soy and edamame which contain polyphenols, resveratrol, isoflavones, genistein are the complex of the protein that contain "KH Good Healthy" cells. US patent 10,195,243 B2, EP patent 3 148 574 B1 and US patent 10,335,446 B2.

We suggest that the mechanism of these complex compounds of natural "KH Good Healthy" proteins which contain good healthy cells which are absorbed into the blood stream to send signal to the body to produce new cells that are healthy. It also sends the RNA signal to the DAMAGED, SICK, AND BAD CELLS that triggers that synthesis of good proteins that transform these cells to become GOOD healthy cells. "KH Good Healthy" proteins also send the RNA signal to the other currently undamaged cells to synthesize good proteins to protect them from being DAMAGED, INFECTED and PRONE to DNA and other cellular alterations.

Besides the above-mentioned mechanism, which we believe are the most important, a secondary or contributing mechanism is the effects of polyphenols, an important component of the grape which contribute to produce "KH Good Healthy" cells. Finally, resveratrol may also be involved, as we know that resveratrol is a naturally occurring stilbenoid derivative found in plants and fruits such as grapes (Vitis vinifera). Resveratrol exhibits potent inhibition against MERS-CoV in vitro and also significantly reduced viral-induced cell death. It is likely that its anti-CoV activity is a result of either activation of cellular survival factors and DNA repair in response to DNA damage via activation of the ERK1/2 signaling pathway or prevention of virus-induced apoptosis via down-regulation of FGF-2 signaling.

RAAS products derive from soy, grapes and rice that contain high concentrations of Apo-A1, Immunoglobulin and Albumin-like proteins. Unlike traditional human plasma derived therapies that limit the product to one single protein, RAAS Nutritionals supplements contain up to 5,055 proteins.

APOA-1 includes HDL, which is a very important protein for a human being. The next important proteins are immunoglobulin and albumin.

RAAS Nutritionals supplements (KUNAMIN®, KHJ®, KHJ-R™ and KUNAKINMIN®) contain up to 5,055 proteins which include 1,299 proteins (of which 959 are newly found proteins found in grapes (Vitis vinifera), 358 proteins (of which 125 are newly found proteins in soybean (Glycine max), 1,223 total proteins (of which 843 are newly found proteins in edamame (Glycine max) and 2,175 proteins (of which 569 are newly found proteins in rice (Oryza sativa).

We have performed an in vitro study by using SDS page to detect the molecular weight of the three main proteins in grape, edamame, soy and rice products that we are looking for: HDL (High Density Lipoprotein) or APOA-1, Immunoglobulin and Albumin.

The in vitro study has shown that these products cover all from the highest molecular weight to the lowest of the protein marker. This proves our analysis of a combination of weight in an SDS page marker.

We used the standard of Human APOA1 lays between 35.0 kDa and 25.0 kDA. Grape, soy and rice APOA1 spreads from 66.2 kDa down to 14.4 kDa, that means all these proteins can be found by SDS page.

Human Immunoglobulin from plasma lays starting at 45.0 kDa and spread down 25.0 kDa. Grape, soy and rice APOA1 spreads from 45.0 kDa down to 14.4 kDa, that means all these proteins can be found by SDS page.

Human albumin which lays between 66.2 kDA and 45.0 kDA. Grape, soy and rice APOA1 spread from 66.2 kDa down to 14.4 kDa, that means all these proteins can be found by SDS page.

For albumin, in addition to the SDS page we used the serum protein electrophoresis that showed the high content of alpha-1, alpha-2 beta and specially gamma (which is immunoglobulin).

For COVID-19 we have no invitro model, therefore we used H1N1 and H3N2 models to evaluate in vitro inhibitory activity of the 24 RAAS Nutritionals test articles against a panel of viruses.

Activity of the articles against IFV. The activity and cytotoxicity results in the influenza virus tests are summarized in Table 5. VX-787 was used as a reference compound. Dose response curves of the test articles in antiviral and cytotoxicity tests. VX-787 showed the expected activities in the tests.

KH 028, Kunamin, KH 024 and KH 019 showed inhibitory activities against influenza H1N1 with EC50 values between 0.028% and 0.092%. KHMC, KunaFlow, KH 029, KH 021 and KHEGW had EC50 values against influenza H1N1 between 0.146% and 0.985%. Kunaking and KHEGY had EC50 values against influenza H1N1 of 1.112% and 2.685%, respectively.

KH 019, KH 028, KH 029, KH 024, Kunamin and KHMC showed inhibitory activities against influenza H3N2 with EC50 values between 0.014% and 0.084%. KunaFlow, Kunaking, KH 021, KHEGW and KHEGY had EC50 values against influenza H3N2 between 0.202% and 1.831%.

For COVID-19 we have no animal model, therefore we used H1N1 model. For in-vivo model we used H1N1 infected mouse model. We have found that APOA-1 from human plasma can prevent and treat H1N1 virus. In our study performed at Wuxi Pharma, one of the top ten CRO's in the world, we found that RAAS-2 (APOA-1) can prevent 100% of the Bird Flu Epidemiology in Mice.

Impressively one-week preventive treatment with 0.2 ml/0.4 ml/mouse iv/ip QD of RAAS-2 (APOA-1) totally protected H1N1-challenged mice from death and body weight loss till the end of this study. The protection of body weight loss by the preventive treatment of RAAS-2 (APOA-1) is even better than that by oseltamivir treatment. However, the therapeutic treatment with 0.2 ml/0.4 ml iv/ip QD of RAAS-2 only protected one mouse out of 5 mice in the group from death and partial body weight loss of all 5 mice days 2 to 5 post H1N1 infection. Other 4 mice in this group died days 4 to 6 post H1N1 infection. In addition, some of the mice in the RAAS-2 therapeutic group (G2) had haematuria day 5 post H1N1 challenge and afterward, indicating that the dose used in this group was beyond mouse tolerance in H1N1 challenge status.

B cells and T cells are the KH good healthy cells to fight back any virus and its mutations just like Omicron. In our in vitro and in vivo studies, we have found that human APOA1 or grape and rice APOA1 will have the ability to fight back lung cancer as well as other kinds of cancers.

We conducted a study at WuXi App Tec titled, Characterization of lymphoid tissues and peripheral blood in nude mouse treated with and without AFCC (Anti Fear of Cancer Cells, a combination of 27 KH human proteins) After whole blood withdrawal, distinct cell lineage was differentiated by cell surface marker proteins. T cells, B cells, activated B cells, mDC, pDC, granulocytes, and monocytes/macrophages were characterized.

AFCC treatment didn't affect CD3+T cell population compared with that in nude mouse with tumor and without tumor. After AFCC treatment, B cell population, on the other hand, increased to the similar percentage as seen in nude mouse no tumor and nude naïve ID: APRON 2020-OK-01 Effect of Kunamin in SARS-CoV-2 RT-PCR Positive Covid-19 Patients [NCT ID not yet assigned] increased with AFCC treatment. Macrophages and granulocytes decreased after AFCC treatment compared with those in nude mouse with tumor. Nude mouse no tumor and nude mouse with AFCC treatment had similar mDC and pDC percentage.

Conclusion: The effect of AFCC on curing tumor through characterizing different cell lineage in lymphoid tissues and peripheral blood in nude mouse was investigated using staining with different marker proteins for distinct cell lineages followed by FACS. T cells, B cells, activated B cells, mDC, pDC, granulocytes, and monocytes/macrophages were characterized in 6 mice.

FACS analysis showed that AFCC treatment had the effect on the population of major cell lineages in immune system. Increased CD3+T cell population was found in nude mouse treated with AFCC compared with that in nude mouse with tumor in spleen and lymph nodes. B cells including activated B cells also increased compared with that in nude mice with tumor in spleen, lymph nodes, and peripheral blood. Granulocytes and macrophages, however, were found to decrease after AFCC treatment in peripheral blood and spleen. Taken together, this study suggests the effect of AFCC on curing tumor through changing the population of major cell lineages in immune system, including spleen, lymph nodes and peripheral blood.

We conducted a study at WuXi App Tec titled, Characterization of draining lymph nodes and peripheral blood in DIO mice treated with KHJ, KH103 and KHGD (KHJ is a grape product, KH103 is a soy product and KHGD Kieu Hoang Gold label) Results summary, the effects of KHJ, KH103 and KHGD on different cell lineages in lymphoid tissues and peripheral blood in DIO mice were investigated by FACS analysis. T cells, B cells, dendritic cells, MDSCs, granulocytes and macrophages were analyzed. Overall, KH103, KHJ and KHGD treatments showed few effects on T cell lineages, macrophages and granulocytes but reduced the percents of B cells in both peripheral blood and draining lymph nodes. They also elevated the percentages of pDCs in blood and reduced the percentages of mDCs in draining lymph nodes. The causes of the alterations remain to be further investigated.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated, mild or moderate pneumonia according to the T.R. Ministry of Health COVID-19 guidelines,
* Adult patients diagnosed with COVID-19
* Being between the age of 18 and 65
* Adult patients diagnosed with COVID-19 by PCR and who have COVID-19 symptoms in CT scan
* Patients who are positive for 2019-nCOVRNA in the test performed on samples taken from the nasopharyngeal area
* Respiratory rate less than 30 / minute
* SpO2 level above 90% in room air
* Finding signs of pneumonia on chest x-ray or tomography
* Having symptoms of COVID19
* Having the skills to understand and approve the informed consent form
* Patients with mild to moderate pneumonia findings according to the above criteria and decided to be treated only in hospital,

Exclusion Criteria:

* Those who are allergic to grape juice and seed extract and / or other drugs and / or excipients of the products included in the standard treatment regimen,
* Pregnant or breastfeeding women
* Those who are not suitable for oral medication
* Patients who have comorbidity and using medication because of their chronic illness
* SpO2 level below 90% in room air
* Those who have diffuse pneumonia findings in chest tomography and radiography
* Patients who are being isolated and treated at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Decrease in COVID-19, cold and flu viral load to become non detected or negative by Polymerase Chain Reaction. | 15 days
  By PCR method.
Produce COVID-19 antibodies | 30 days
  Produce COVID-19 antibodies from 0 au/mL up to >10.0 aU/mL. Chemiluminescent microparticle immunoassay (CMIA)
Decrease in bacteria microbe load to become non detected or reduced. | 30 days
  Reverse transcriptase polymerase chain reaction (TaqManqPCR)
Normalization of fever, respiratory rate, oxygen saturation and alleviation of cough. | 15 days
  Clinical recovery time (normalization of fever, respiratory rate and oxygen saturation and alleviation of cough). NEWS2 Scoring system
Changes in hospitalization / recovery time, discharge from hospital | 30 days
  Hospital records
Improvement in coronavirus symptoms including ferritin, d-dimer, CRP, lymphocyte count. | 30 days
  Comprehensive metabolic panel (CMP)

SECONDARY OUTCOMES:
Reduction of diabetes blood sugar level | 30 days
  Comprehensive metabolic panel (CMP)
Increase HDL decrease LDL and triglycerides | 30 days
  Comprehensive metabolic panel (CMP)

CONTACTS AND LOCATIONS:
Overall Officials: Kieu Hoang, Study Chair — RAAS Nutritionals, LLC
Locations (1):
- Kayseri City Hospital, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No